CLINICAL TRIAL: NCT02322710
Title: Multicentre, Randomized, Parallel Group, Non-inferiority, Open-label Study Aiming at Comparing the Healing Rates (With Blinded Assessment Based on Photographs) of TULLEGRAS M.S.® With URGOTUL® in the Treatment of Surgical Acute Wounds.
Brief Title: Comparison of Efficacy on Healing, and Safety of Two Dressings Urgotul and TulleGras MS on Surgical Acute Wounds.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Fovea (Other)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LINE4002; 2014-A00914-43 (Other: ANSM (French Health Agency) Registry number for biomedical research)
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2017-03

CONDITIONS: Surgical Acute Wounds
Keywords: non-inferiority; randomized; TulleGras; Urgotul; healing; surgical acute wounds; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TulleGras M.S. (Active Comparator): Sterile dressing that consists of viscose tissue coated with mineral vaseline
  Interventions: Device: TulleGras M.S.: Vaseline gauze
- Urgotul (Active Comparator): Sterile, hydrocolloid dressing, that consists of a polyester fabric coated with hydrocolloid particles and vaseline
  Interventions: Device: Urgotul: Low-adherent dressing

INTERVENTIONS:
Device: Urgotul: Low-adherent dressing
  Arms: Urgotul
Device: TulleGras M.S.: Vaseline gauze
  Arms: TulleGras M.S.

SUMMARY:
Evaluation of non-inferiority on healing rates of two dressings Urgotul and TulleGras MS in the treatment of surgical acute wounds.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject.
* Aged 18 to 75 years
* With a planned surgery:
* Of abdominal location
* Leading to an acute wound of a maximum total length ≤ 18 cm (corresponding to 2 investigational products)
* Absence of clinical sign suggestive of worsened wound (assessed only at the randomization visit)
* Followed-up in surgery department
* Written and signed informed consent obtained
* Affiliated to the French Social Security system or equivalent.

Exclusion Criteria:

* Underlying pathology that may interfere with wound healing in the opinion of the Investigator (human immunodeficiency virus [HIV], cancer, immunodeficiency disease, generalized infection, systemic disease ...). The presence of low-risk prostate cancer according to the Amico classification (1) (PSA<10 ng/mL and Gleason's score < 6 and clinical grade T1c ou T2a) or a grade T1 (a or b) N0M0 renal cancer which requires surgery without adjuvant therapy (radiotherapy, chemotherapy, hormonal therapy...), in a patient whose general condition is preserved without significant comorbidity or signs of malnutrition are not considered as a non- inclusion criteria
* Inadequately controlled diabetes (Glycosylated hemoglobin > 8%)
* Hypo or hyperthyroidism
* Intake of a systemic treatment with glucocorticoids or immunosuppressives
* Known allergy to one of study dressings components
* Participation in a clinical trial in the month prior to his/her inclusion in the study
* Pregnancy or breastfeeding or of childbearing potential and saying not to use contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger LESAUNIER, MD, Study Director — Mylan
Locations (33):
- France (33):
  - Research facility ID ORG-001264, Ajaccio
  - Research facility ID ORG-001263, Angoulême
  - Research facility ORG-001090, Athis-Mons
  - Research facility ORG-001101, Aubervilliers
  - Research facility ID ORG-001099, Carpentras
  - Research facility ORG-001099, Carpentras
  - Research facility ORG-001107, Cornebarrieu
  - Research facility ID ORG-001223, La Rochelle
  - Research facility ORG-001096, Levallois-Perret
  - Research facility ID ORG-001276, Lille
  - Research facility ORG-001102, Lille
  - Research facility ORG-001360, Lyon
  - Research facility ORG-001132, Mantes-la-Jolie
  - Research facility ID ORG-001133, Montpellier
  - Research facility ORG-001133, Montpellier
  - Research facility ID ORG-001220, Montreuil
  - Research facility ID ORG-001189, Nice
  - Research facility ID ORG-001190, Ollioules
  - Research facility ID ORG-001088, Paris
  - Research facility ID ORG-001105, Paris
  - Research facility ORG-001105, Paris
  - Research facility ID ORG-001134, Paris
  - Research facility ID ORG-001265, Paris
  - Research facility ORG-001088, Paris
  - Research facility ID ORG-001221, Paris
  - Research facility ORG-001166, Pierre-Bénite
  - Research facility ID ORG-001278, Reims
  - Research facility ORG-001137, Roubaix
  - Research facility ORG-001136, Rouen
  - Research facility ORG-001089, Saint-Nazaire
  - Research facility ID ORG-001222, Sarreguemines
  - Research facility ORG-001097, Sarreguemines
  - Research facility ORG-001093, Toulon

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 patients were not randomized Presence of clinical sign suggestive of worsened wound assessed at the randomization visit (n=4)
Groups:
- TulleGras M.S.: Sterile dressing that consists of viscose tissue coated with mineral vaseline
  TulleGras M.S.: Vaseline gauze
- Urgotul: Sterile, hydrocolloid dressing, that consists of a polyester fabric coated with hydrocolloid particles and vaseline
  Urgotul: Low-adherent dressing
Period: Overall Study
Arm/Group | TulleGras M.S. | Urgotul
Started (Patients randomized) | 105 | 99
Safety Population | 105 | 99
Full Analysis Population (No efficacy assessment post-baseline (N=1)) | 105 | 98
Completed (Per protocol population) | 85 | 73
Not Completed | 20 | 26
Not completed — No efficacy assessment post-baseline | 0 | 1
Not completed — Protocol Violation | 20 | 25

BASELINE CHARACTERISTICS:
Population: Full analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | TulleGras M.S. | Urgotul | Total
Number analyzed (Participants) | 105 | 98 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Full analysis population = 203
  years | 52.4 (13.2) | 54.4 (14.1) | 53.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full analysis population = 203
  Participants
    Female | 39 | 43 | 82
    Male | 66 | 55 | 121
Weight [Mean (Standard Deviation); unit: Kg] — Population: Full analysis population = 203 Missing data = 10
  Kg
    number analyzed (Participants) | 99 | 94 | 193
    (all) | 85.4 (21.6) | 83.0 (18.9) | 84.2 (20.3)
Height [Mean (Standard Deviation); unit: Cm] — Population: Full analysis population = 203 Missing data = 10
  Cm
    number analyzed (Participants) | 99 | 94 | 193
    (all) | 170.4 (9.6) | 170.0 (9.2) | 170.2 (9.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] — Population: Full analysis population = 10 Missing data = 10
  kg/m²
    number analyzed (Participants) | 99 | 94 | 193
    (all) | 29.6 (8.3) | 28.9 (7.2) | 29.2 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Healing (100% of Epithelialization).
Description: Using photographs,independent assessor blinded assessment.
Time Frame: Day 21
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | TulleGras M.S. | Urgotul
Number analyzed (Participants) | 85 | 73
Participants | 77 | 67
Statistical Analysis 1: Comparison: TulleGras M.S. vs Urgotul; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper limit of the 95% confidence interval of the observed difference between healing rates at D21 (Urgotul® - Tullegras M.S.®) in the PP population did not exceed +10%; Difference in Percentages = 1.2, 97.5% CI 1-sided [upper limit 10.0], Standard Deviation 4.5

ADVERSE EVENTS:
Arm/Group | TulleGras M.S. | Urgotul
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/99
Serious Adverse Events (participants affected / at risk) | 14/105 | 7/99
Other Adverse Events (participants affected / at risk) | 23/105 | 30/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TulleGras M.S. (N=105) | Urgotul (N=99)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
gastric fistula (Gastrointestinal disorders) | 1 | 0
eschereschia coli (Infections and infestations) | 1 | 1
pyelonephretis (Infections and infestations) | 0 | 2
hyperthermia (General disorders) | 1 | 1
post procédural constipation (Injury, poisoning and procedural complications) | 1 | 0
dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
haemorroids thrombosed (Vascular disorders) | 1 | 0
anaemia (Blood and lymphatic system disorders) | 2 | 0
urinary retention (Renal and urinary disorders) | 1 | 1
hypokaliaemia (Investigations) | 1 | 0
lymphopenia (Blood and lymphatic system disorders) | 1 | 0
ileus (Gastrointestinal disorders) | 0 | 1
hypertension (Vascular disorders) | 0 | 1
prostate sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
asymptomatic cholostasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TulleGras M.S. (N=105) | Urgotul (N=99)
procedural pain (Injury, poisoning and procedural complications) | 9 | 13
abdominal pain (Gastrointestinal disorders) | 10 | 2
nausea (Gastrointestinal disorders) | 1 | 9
pain (General disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No